CLINICAL TRIAL: NCT02862106
Title: Second Stage:Open-label Study of Therapeutic Hepatitis B Vaccine (Mimogen-based) in Treating Chronic Hepatitis B Patients
Brief Title: Second Stage:Open-label Study of Therapeutic Hepatitis B Vaccine (Mimogen-based) for Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing Jiachen Biotechnology Ltd. (Industry)
Collaborators: Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 71006.01-2
Record Dates: First submitted 2016-08-06; First posted 2016-08-10 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2016-11

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; HBeAg positive; Therapeutic HBV Vaccine; HBV-specific Cytotoxic T Lymphocyte
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- εPA-44 900μg group-placebo (Experimental): These subjects from the placebo group of protocol 71006.01 InjectεPA-44 900μg at week 83,86,89,92,95,98,101,104,108,112,116,120,124,128
  Interventions: Biological: εPA-44
- εPA-44 900μg group-εPA-44 600μg (Experimental): These subjects from the εPA-44 600μg group of protocol 71006.01 Inject εPA-44 900μg at week 83,86,89,92,95,98,101,104,108,112,116,120,124,128
  Interventions: Biological: εPA-44
- εPA-44 900μg group-εPA-44 900μg (Experimental): These subjects from the εPA-44 900μg group of protocol 71006.01 Inject εPA-44 900μg at week 83,86,89,92,95,98,101,104,108,112,116,120,124,128
  Interventions: Biological: εPA-44
- Follow-up group-placebo (No Intervention): These subjects from the placebo group of protocol 71006.01 Do not give any intervention, follow-up observation only
- Follow-up group-εPA-44 600μg (No Intervention): These subjects from the εPA-44 600μg group of protocol 71006.01 Do not give any intervention, follow-up observation only
- Follow-up group-εPA-44 900μg (No Intervention): These subjects from the εPA-44 900μg group of protocol 71006.01 Do not give any intervention, follow-up observation only

INTERVENTIONS:
Biological: εPA-44 — subcutaneously injection of εPA-44 900μg at week 83,86,89,92,95,98,101,104,108,112,116,120,124,128
  Other Names: Therapeutic HBV vaccine
  Arms: εPA-44 900μg group-placebo; εPA-44 900μg group-εPA-44 600μg; εPA-44 900μg group-εPA-44 900μg

SUMMARY:
The purpose is to evaluate efficacy and safety of therapeutic HBV vaccine (mimogen-based) treatment in chronic hepatitis B patients and to explore the most effective dosage and provide the rational for optimal dosing schedule.

DETAILED DESCRIPTION:
Second stage(76-144 weeks):

In this follow-up stage the trial is open designed, and all the subjects completed the first stage study(0-76 weeks)

1. Subjects with virological response but no serological response/with serological response but no virological response/neither virological nor serological response in the first stage, and be willing to continue the this follow-up study, will be treated by εPA-44 900 μg at week 80,83,86,89,92,95,98,101,104,108,112,116,120,124,128.
2. Subjects with both virological and serological response, will be followed-up to 144 weeks with no Adefovir Dipivoxil or εPA-44 900 μg treatment.

The definition of response as below:

1. Virological response: HBV DNA<2.93×10∧3IU/ml at 76 weeks;
2. Serological response: serological conversion of HBeAg at 76 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects completed the first stage study(0-76 weeks) and willing to willing to participate in the trial
2. Uses effective contraception for subject with child-bearing potential (including females and female partners of males)
3. Understands and signs ICF approved by EC
4. Willing to comply with the study procedures and complete the study

Exclusion Criteria:

1.Any other factors inappropriate for enrollment in the study or study completion in the view of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wei, Ph.D., Principal Investigator — Hepatitis Institute of Peking University People's Hospital
Locations (9):
- China (9):
  - Renmin Hosptial of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - 81th Hospital of PLA, Nanjing, Jiangsu
  - TangDu Hospital, XiAn, Shanxi
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - 302 Militray Hosptial of China, Beijing
  - Hepatitis Institute of Peking University People's Hospital, Beijing
  - Southwest Hospital, Chongqing

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants completed the first stage(0-76weeks),enrolled at 9 sites in the China. The first participant was screened on 19 November 2011.
Pre-assignment Details: 209 participants entered the second stage of the study , and comprise the Safety Analysis Set and the Full Analysis Set
Groups:
- εPA-44 900μg: Inject εPA-44 900μg at week 83,86,89,92,95,98,101,104,108,112,116,120,124,128
  εPA-44: Inject εPA-44 900μg at week 83,86,89,92,95,98,101,104,108,112,116,120,124,128
- Follow-up Group: Do not give any intervention, follow-up observation only
Period: Overall Study
Arm/Group | εPA-44 900μg | Follow-up Group
Started | 183 | 26
Completed | 145 | 20
Not Completed | 38 | 6
Not completed — Adverse Event | 4 | 0
Not completed — Protocol Violation | 16 | 1
Not completed — Lost to Follow-up | 15 | 5
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Subjects moved to other city | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population
Groups:
- εPA-44 900μg Group-placebo: These subjects from the placebo group of protocol 71006.01 Inject εPA-44 900μg at week 83,86,89,92,95,98,101,104,108,112,116,120,124,128
- Total: Total of all reporting groups
Arm/Group | Follow-up Group-placebo | Follow-up Group-εPA-44 600μg | Follow-up Group-εPA-44 900μg | εPA-44 900μg Group-placebo | εPA-44 900μg Group-εPA-44 600μg | εPA-44 900μg Group-εPA-44 900μg | Total
Number analyzed (Participants) | 3 | 12 | 10 | 64 | 56 | 58 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 12 | 10 | 64 | 56 | 58 | 203
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (6.03) | 25.2 (4.39) | 25.8 (8.02) | 30.4 (7.56) | 29.6 (9.14) | 29.4 (7.61) | 29.4 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 3 | 16 | 8 | 16 | 50
  Male | 2 | 6 | 7 | 48 | 48 | 42 | 153
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.69 (4.043) | 21.23 (2.181) | 21.42 (2.601) | 21.95 (2.615) | 21.76 (3.273) | 22.12 (2.792) | 21.89 (2.835)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients About HBeAg / Anti-HBe Seroconversion at the End of the Follow-up Period
Description: Primary endpoint data were summarised under "End of Study",using the last available post-baseline observation(Last Observation Carried Forward,LOCF)
Time Frame: Endpoint (LOCF), up to 144 weeks
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Groups:
- εPA-44 900μg Group-placebo; εPA-44 900μg Group-εPA-44 600μg: These subjects from the εPA-44 600μg group of protocol 71006.01 Inject εPA-44 900μg at week 83,86,89,92,95,98,101,104,108,112,116,120,124,128
Arm/Group | Follow-up Group-placebo | Follow-up Group-εPA-44 600μg | Follow-up Group-εPA-44 900μg | εPA-44 900μg Group-placebo | εPA-44 900μg Group-εPA-44 600μg | εPA-44 900μg Group-εPA-44 900μg
Number analyzed (Participants) | 3 | 11 | 9 | 62 | 55 | 58
percentage of participants | 66.7 | 100 | 100 | 38.7 | 40 | 34.5

2. Secondary Outcome: The Proportion of Patients About HBeAg / Anti-HBe Seroconversion at week95,108,120,144
Time Frame: week95,108,120,144
Population: Intention to treat population
Measure: Number; unit: percentage of paricipant
Arm/Group | Follow-up Group-placebo | Follow-up Group-εPA-44 600μg | Follow-up Group-εPA-44 900μg | εPA-44 900μg Group-placebo | εPA-44 900μg Group-εPA-44 600μg | εPA-44 900μg Group-εPA-44 900μg
Number analyzed (Participants) | 3 | 11 | 9 | 62 | 55 | 58
percentage of paricipant
  Week 95 | 66.7 | 100 | 100 | 25.8 | 21.8 | 34.5
  Week 108 | 33.3 | 100 | 55.6 | 32.3 | 32.7 | 34.5
  Week 120 | 33.3 | 72.7 | 44.4 | 29.0 | 30.9 | 25.9
  Week 144 | 33.3 | 81.8 | 100 | 37.1 | 32.7 | 27.6

3. Secondary Outcome: The Proportion of Patients With Both Negative HBeAg and HBeAb.
Time Frame: week95,108,120,144
Population: intention to treat population
Measure: Number; unit: percentage of paricipants
Arm/Group | Follow-up Group-placebo | Follow-up Group-εPA-44 600μg | Follow-up Group-εPA-44 900μg | εPA-44 900μg Group-placebo | εPA-44 900μg Group-εPA-44 600μg | εPA-44 900μg Group-εPA-44 900μg
Number analyzed (Participants) | 3 | 11 | 9 | 62 | 55 | 58
percentage of paricipants
  Week 95 | 33.3 | 0 | 0 | 1.6 | 0 | 1.7
  Week 108 | 33.3 | 0 | 0 | 3.2 | 3.6 | 1.7
  Week 120 | 0 | 0 | 0 | 4.8 | 0 | 3.4
  Week 144 | 33.3 | 0 | 0 | 4.8 | 3.6 | 6.9

4. Secondary Outcome: The Proportion of Patients About HBsAg / Anti-HBs Seroconversion at Week 95,108,120,144
Time Frame: week95,108,120,144
Population: intention to treat population
Measure: Number; unit: percentage of participants
Groups:
- εPA-44 900μg Group-εPA-44 600μg: These subjects from theεPA-44 600μg group of protocol 71006.01 Inject εPA-44 900μg at week 83,86,89,92,95,98,101,104,108,112,116,120,124,128
Arm/Group | Follow-up Group-placebo | Follow-up Group-εPA-44 600μg | Follow-up Group-εPA-44 900μg | εPA-44 900μg Group-placebo | εPA-44 900μg Group-εPA-44 600μg | εPA-44 900μg Group-εPA-44 900μg
Number analyzed (Participants) | 3 | 11 | 9 | 62 | 55 | 58
percentage of participants
  Week 95 | 0 | 0 | 0 | 0 | 0 | 0
  Week 108 | 0 | 0 | 0 | 0 | 0 | 0
  Week 120 | 0 | 0 | 0 | 0 | 0 | 0
  Week 144 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: The Proportion of Patients With Both Negative HBsAg and HBsAb.
Time Frame: week95,108,120,144
Population: intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Follow-up Group-placebo | Follow-up Group-εPA-44 600μg | Follow-up Group-εPA-44 900μg | εPA-44 900μg Group-placebo | εPA-44 900μg Group-εPA-44 600μg | εPA-44 900μg Group-εPA-44 900μg
Number analyzed (Participants) | 3 | 11 | 9 | 62 | 55 | 58
percentage of participants
  Week 95 | 0 | 0 | 0 | 0 | 0 | 0
  Week 108 | 0 | 0 | 0 | 0 | 0 | 0
  Week 120 | 0 | 0 | 0 | 0 | 0 | 0
  Week 144 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: The Proportion of Patients With HBV DNA Levels Undetectable or Below the Detection Limit
Time Frame: week95,108,120,144
Population: intention to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Follow-up Group-placebo | Follow-up Group-εPA-44 600μg | Follow-up Group-εPA-44 900μg | εPA-44 900μg Group-placebo | εPA-44 900μg Group-εPA-44 600μg | εPA-44 900μg Group-εPA-44 900μg
Number analyzed (Participants) | 3 | 11 | 9 | 62 | 55 | 58
percentage of participants
  Week 95 | 100 | 90.9 | 100 | 25.8 | 30.9 | 36.2
  Week 108 | 66.7 | 90.9 | 55.6 | 33.9 | 25.5 | 34.5
  Week 120 | 33.3 | 63.6 | 44.4 | 32.3 | 23.6 | 29.3
  Week 144 | 66.7 | 63.6 | 100 | 35.5 | 30.9 | 39.7

7. Secondary Outcome: Change From Baseline by Visit for Serum HBV DNA
Time Frame: week95,108,120,144
Population: intention to treat population
Measure: Mean (Standard Deviation); unit: log_10 IU/mL
Arm/Group | Follow-up Group-placebo | Follow-up Group-εPA-44 600μg | Follow-up Group-εPA-44 900μg | εPA-44 900μg Group-placebo | εPA-44 900μg Group-εPA-44 600μg | εPA-44 900μg Group-εPA-44 900μg
Number analyzed (Participants) | 3 | 11 | 9 | 62 | 55 | 58
log_10 IU/mL
  Baseline values of log | 8.1 (0.64) | 7.6 (0.97) | 7.5 (1.1) | 7.8 (0.88) | 8.1 (0.9) | 8.0 (0.99)
  Week 95 decreases from baseline | 6.0 (0.67) | 5.1 (1.23) | 5.6 (0.92) | 2.8 (1.83) | 2.7 (2.18) | 2.9 (2.34)
  week 108 decreases from baseline | 6.3 (0.14) | 5.2 (1.24) | 5.4 (0.71) | 3.0 (2.10) | 3.1 (2.17) | 3.2 (2.40)
  week 120 decreases from baseline | 5.5 (0.97) | 5.2 (0.99) | 5.9 (0.83) | 3.0 (2.19) | 3.3 (1.94) | 2.8 (2.66)
  week 144 decreases from baseline | 5.6 (0.34) | 5.1 (1.09) | 5.6 (1.21) | 3.2 (2.27) | 4.1 (1.77) | 3.3 (2.69)

8. Secondary Outcome: Percentage of Participants Who Achieved HBV DNA Levels <29300 IU/mL or HBV DNA Load Decrease Equal or Greater Than 2 Log Scales;
Time Frame: week95,108,120,144
Population: intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Follow-up Group-placebo | Follow-up Group-εPA-44 600μg | Follow-up Group-εPA-44 900μg | εPA-44 900μg Group-placebo | εPA-44 900μg Group-εPA-44 600μg | εPA-44 900μg Group-εPA-44 900μg
Number analyzed (Participants) | 3 | 11 | 9 | 62 | 55 | 58
percentage of participants
  Week 95 | 100 | 100 | 100 | 59.7 | 52.7 | 60.3
  Week 108 | 66.7 | 100 | 55.6 | 61.3 | 60.0 | 60.3
  Week 120 | 66.7 | 72.7 | 44.4 | 54.8 | 58.2 | 43.1
  Week 144 | 66.7 | 81.8 | 100 | 61.2 | 58.2 | 55.2

9. Secondary Outcome: Change From Baseline by Vsit for HBeAg Titer.
Description: Measuring the change in value of each visit viewpoints HBeAg titers decreased compared with baseline values
Time Frame: week95,108,120,144
Population: intend to treat population
Measure: Mean (Standard Deviation); unit: IU/ML
Arm/Group | Follow-up Group-placebo | Follow-up Group-εPA-44 600μg | Follow-up Group-εPA-44 900μg | εPA-44 900μg Group-placebo | εPA-44 900μg Group-εPA-44 600μg | εPA-44 900μg Group-εPA-44 900μg
Number analyzed (Participants) | 3 | 11 | 9 | 62 | 55 | 58
IU/ML
  baseline of HBeAg titers | 1276.5 (1447.33) | 758.5 (1287.52) | 285.9 (411.9) | 681.9 (658.52) | 958.3 (929.45) | 880.9 (1368.65)
  Week 95 decreases from baseline | -1276.3 (1447.33) | -758.3 (1287.52) | -285.7 (411.9) | -435.8 (685.25) | -617.1 (913.09) | -550.7 (1834.16)
  week 108 decreases from baseline | -446.3 (237.59) | -758.3 (1287.52) | -38.9 (49.73) | -476.8 (728.21) | -807.0 (1011.18) | -602.9 (1755.50)
  week 120 decreases from baseline | -446.3 (237.64) | -979.9 (1463.54) | -314.4 (576.36) | -500.7 (654.06) | -769.4 (1017.49) | -486.3 (927.24)
  week 144 decreases from baseline | -446.3 (237.59) | -923.9 (1379.30) | -285.7 (411.9) | -546.3 (629.66) | -788.4 (887.7) | -691.5 (1708.44)

ADVERSE EVENTS:
Groups:
- Follow-up Group: Do not give any intervention, follow-up observation only All safety analyzes were analyzed in a safe population, and since 1 subjects had no safety data, they were excluded from the safety population
- εPA-44 900μg Group: Inject εPA-44 900μg at week 83,86,89,92,95,98,101,104,108,112,116,120,124,128 All safety analyzes were analyzed in a safe population, and since 5 subjects had no safety data, they were excluded from the safety population
Arm/Group | Follow-up Group | εPA-44 900μg Group
Serious Adverse Events (participants affected / at risk) | 0/25 | 5/178
Other Adverse Events (participants affected / at risk) | 2/25 | 43/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Follow-up Group (N=25) | εPA-44 900μg Group (N=178)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Severe chronic hepatitis B (Infections and infestations) | 0 (0) | 2 (2)
Acute exacerbation of Chronic hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Follow-up Group (N=25) | εPA-44 900μg Group (N=178)
Injection site pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Injection site swelling (Skin and subcutaneous tissue disorders) | 0 | 2
Injection site erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 8
Nasopharyngitis (Infections and infestations) | 1 | 5
weakness (General disorders) | 0 | 3
fever (General disorders) | 1 | 1
ALT increased (General disorders) | 0 | 3
AST increased (Investigations) | 0 | 2
Leukocytes in urine positive (Investigations) | 0 | 2
Elevated transaminase (Investigations) | 0 | 2
insomnia (Nervous system disorders) | 0 | 2
Mouth ulcers (Gastrointestinal disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 3
Gum pain (Gastrointestinal disorders) | 0 | 2
Gingival swelling (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators can't publish articles relevant to the study unless the sponsor permits.